CLINICAL TRIAL: NCT06968182
Title: The Effect of Sodium on Erythrocyte Salt Sensitivity, Syndecan-1 and Heparin Sulfate in Healthy Subjects: A Randomized, Double-Blinded, Placebo-Controlled, Cross-Over Study
Brief Title: The Effect of Sodium on Erythrocyte Salt Sensitivity, Syndecan-1 and Heparin Sulfate in Healthy Subjects.
Acronym: EGNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frank Mose (Other)
Collaborators: Region MidtJylland Denmark (Other)
Responsible Party: Sponsor-Investigator, Frank Mose, Clinical Professor, Md. Ph.d., Region MidtJylland Denmark
Organization: Region MidtJylland Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: RLS-1-2015; 1-10-72-351-15 (Other: De Videnskabsetiske Komiteer For Region Midtjylland)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sodium; Renal Function; Blood Pressure
Keywords: sodium; Renal Handling
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Design The study was conducted as a randomized, double-blinded, placebo-controlled, crossover trial. Subjects received a four days standardized and sodium reduced diet and NaCl tablets or placebo in random order. Each treatment period was followed by an examination day. The examination days were separated by a wash-out period of at least three weeks.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High sodium (Active Comparator): During the high sodium period, the subjects received 200 mmol sodium in tablets. The standardized sodium reduced diet contained 100 mmol sodium.
  Interventions: Dietary Supplement: Sodium Chloride
- Low sodium (Placebo Comparator): During the low sodium period, the subjects received the placebo tablets contained 86 mg of potato starch and 85 mg lactose monohydrate. The standardized sodium reduced diet contained 100 mmol sodium.
  Interventions: Dietary Supplement: Sodium Chloride

INTERVENTIONS:
Dietary Supplement: Sodium Chloride — During the examination day after a baseline period, from 11.00 AM to 11.30 AM, a sustained infusion of 1 L isotonic NaCl, was administered.

SUMMARY:
The study was a double-blinded, randomized, placebo-controlled cross-over study. 27 healthy subjects received a four days standardized, sodium reduced diet (100 mmol sodium) and treatment with sodium chloride (200 mmol sodium) or placebo in a randomized order. After the treatment the subjects went to an examination day. With 1 L isotonic sodium chlorid intravenous in 25 minutes, the subjects were further sodium and volume loaded. Change in salt blood test (SaBT), syndecan-1(syn-1) and heparan sulfate (HS), brachial and central blood pressure (BP), pulse wave velocity (PWV) and augmentation index (AIx) were measured. Baseline blood samples were taken before the treatment periods

DETAILED DESCRIPTION:
Background: The endothelium is lined with endothelial glycocalyx (EG). EG protects the endothelium and functions as a barrier between blood and endothelium. Due to negative charges EG has a strong ability to buffer sodium. In vitro studies indicate that sodium overload can damage the EG and reduce the sodium buffer capacity. This could cause endothelial dysfunction and might lead to cardiovascular disease. EG can be measured by the erythrocyte salt sensitivity (ESS) and shedding of glycocalyx.

Purpose: The investigators aimed to examine the effect of dietary sodium balance on EG in healthy subjects.

Methods: In a double blinded, randomized, placebo controlled cross over study, 27 healthy subjects received a four days sodium reduced diet and treatment with NaCl or placebo in randomized order. Afterwards the subjects were further sodium and volume loaded with 1 L isotonic NaCl intravenously. Changes in ESS and blood pressure were measured.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age 18-50 years,
* BMI 18.5-30.0 kg/m2,
* Signed concent.
* Fertile women with safe contraception during the whole examination period.

Exclusion Criteria:

* Alcohol consumption > 7 drinks per week for women and, > 14 drinks per week for men.
* Smoking,
* Substance abuse
* Current use of medicine except contraception,
* Office BP > 140/90
* History or signs of clinically relevant kidney, heart, liver, lung, neurological, or endocrine diseases, neoplastic disorders,
* Pregnancy or lactation
* Blood donation within 1 month of the first investigation,
* Clinically relevant abnormal blood/urine sample or electrocardiography.

Withdrawal criteria:

* Development of exclusion criteria
* Suspicion of poor compliance to study medication
* Withdrawal of signed concent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
erythrocyte salt sensitivity (ESS) | From enrollment and at the end of the second examination day, aprox. 3-4 months
  eGC is in dynamic equilibrium between biosynthesis of new components and release of "old". This is called shedding and the protein components can be measured in the plasma. Shedding is increased in e.g. sepsis, ischemia, kidney failure and severe bleeding {{38 Mulivor,A.W. 2004; 36 Salmon, Andrew H J AH 2012; 48 Sillesen,M. 2014; 49 Nelson,A. 2008; 50 Steppan,J. 2011}}{{35 Nieuwdorp,M. 2005}}.
  The erythrocytes (RBC) also posses a glycocalyx-layer. Intact glycocalyx of both endothelium and erythrocytes is important for maintenance of electrostatic forces and frictionless passage of the RBC through the capillaries{{20 Oberleithner,H. 2013; 26 Oberleithner,H. 2012; 7 Oberleithner,H. 2015}} Deterioration of eGC affect the RBC, and the surface of the RBC becomes a mirror image of the properties of eGC{{20 Oberleithner,H. 2013; 8 Oberleithner,H. 2014}}.
  Change in the RBC membrane can be demonstrated by a "salt-blood test-mini"{{18 Oberleithner,H. 2013; 99 Oberleithner,H. 2016}}. This is an

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N. Bech, professor, Study Director — University Clinic in Nephrology and Hypertension, Gødstrup Hospital, Hospitalsparken 15, 7400 Herning, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ostergaard AM, Sonderbaek RL, Vrist MH, Rosenbaek JB, Mose FH, Bech JN. Effect of sodium balance on levels of nitrates in healthy subjects: Posthoc analysis of a randomized, double-blinded, placebo-controlled, crossover study. Physiol Rep. 2025 Aug;13(16):e70512. doi: 10.14814/phy2.70512. PMID 40827100